CLINICAL TRIAL: NCT07405775
Title: SleepFix for Youth: Digital Behavioural Therapy for Insomnia With E-Psychologist Support
Acronym: iSLEEPY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Woolcock Institute of Medical Research (Other)
Collaborators: Macquarie University, Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025/ETH19111
Record Dates: First submitted 2025-11-24; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-08

CONDITIONS: Insomnia
Keywords: young people; adolescents; insomnia; CBTi; digital behavioural therapy for insomnia; sleep restriction therapy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Masking Description: The research staff, e-psychologist and Principle Chief Investigator will not be blinded to the study as they will be managing the online study directly which will lend itself to knowing which groups participants are allocated to. Participants will not be blinded as they will know what treatment they receive.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment: SleepFix + e-psychologist support calls (Experimental): Participants receive the SleepFix mobile application with weekly support calls from an e-psychologist for 3 weeks, with an optional additional 3 weeks of use. SleepFix will deliver digital brief behavioural therapy for insomnia (dBBTi) based on sleep consolidation therapy. The program aims to improve sleep efficiency by tailoring a personalised sleep window and gradually adjusting it. Participants will be instructed to use SleepFix for a 3-week period, with the option to continue for up to an additional 3 weeks. Weekly 15-20 minute sleep support calls from a trained e-psychologist will provide guidance, troubleshooting, and encouragement throughout the intervention period. Participants will also receive access to educational videos on sleep retraining.
  Interventions: Behavioral: SleepFix + e-psychologist support calls
- Sleep Health Education (Active Control) (Active Comparator): Participants randomised to this arm will receive three online sleep health education modules delivered via email every two weeks over a 6-week period. The modules provide information on sleep and healthy sleep habits. Control group participants will be offered full access to the SleepFix application with the weekly support calls from an e-psychologist after completing their final follow-up assessment at week 14.
  Interventions: Behavioral: Sleep Health Education (Active control)

INTERVENTIONS:
Behavioral: SleepFix + e-psychologist support calls — SleepFix mobile application uses Sleep Retraining Therapy (SRT) which aims to reduce excess time spent in bed awake and reset sleep by matching time in bed to total sleep time (TST). There are four stages to the SleepFix app and participants will progress based on completion of each stage. Participants are required to enter sleep and bedtime/wake data into the smartphone app for baseline referencing and determination of sleep therapy. SleepFix uses an algorithm that calculates optimal sleep efficiency based on participants data
  Other Names: sleep restriction therapy; sleep consolidation therapy; sleep retraining therapy
  Arms: Treatment: SleepFix + e-psychologist support calls
Behavioral: Sleep Health Education (Active control) — Three online sleep health education modules are provided to participants. It included information about healthy sleep, insomnia, sleep hygiene practices and information on general strategies for managing sleep for insomnia.
  Other Names: sleep education
  Arms: Sleep Health Education (Active Control)

SUMMARY:
This pilot randomised, open-label, parallel-group controlled trial will evaluate the feasibility, acceptability and effects of a psychologist-supported digital behavioural therapy for insomnia (dBTi) compared to a wait-listed active control (digital sleep health education) in young people aged 16-24 years with insomnia symptoms.

The primary objectives are to evaluate the feasibility of conducting a full-scale trial by assessing recruitment, consent and randomisation rates, intervention uptake, and data completeness. Secondary objectives include exploring treatment effects on insomnia severity (Insomnia Severity Index), sleep diary metrics, sleep quality, fatigue, and mood (depression and anxiety symptoms). Post-intervention interviews will assess participant experience and acceptability.

Results will inform the design of a larger randomised controlled trial.

DETAILED DESCRIPTION:
Insomnia is a common sleep disorder among young people, with significant impacts on mental health, daily functioning, and wellbeing. Cognitive Behavioural Therapy for Insomnia (CBTi) is the recommended first-line treatment, and digital delivery offers a scalable way to improve access. Despite strong evidence in the adult literature supporting digital CBTi and standalone individual treatment components of CBTi (e.g., sleep restriction), there is limited research examining their effectiveness and feasibility in young populations.

This pilot, open-label, parallel-group randomised controlled trial will evaluate the feasibility, acceptability, and effects of SleepFix, a smartphone application delivering digital Brief Behavioural Therapy for Insomnia (dBBTi), supported by weekly contact with an e-psychologist, compared to an active control consisting of online Sleep Health Education modules.

Participants (n = 40) aged 16-24 years with insomnia symptoms will be recruited nationally via online advertisements and community networks. Following online pre-screening and a telephone eligibility interview, eligible participants will provide electronic consent and complete baseline questionnaires and a 7-day sleep diary before randomisation (1:1) to one of two groups:

1. Intervention group: Participants will use the SleepFix mobile app, which delivers digital Brief Behavioural Therapy for Insomnia (based primarily on sleep restriction therapy), alongside weekly 15-20minute calls from an e-psychologist for 3 weeks, with an optional additional 3 weeks of therapy.
2. Control group: Participants will receive three online Sleep Health Education modules delivered bi-weekly across a 6-week period. After completing the final follow-up, participants in the control group will be offered access to the SleepFix app and e-psychologist support.

Assessments will occur at baseline, 6 weeks (post-treatment), and 14 weeks (follow-up). The primary outcomes are feasibility measures, including recruitment, consent and randomisation rates, intervention uptake, and data completion. Secondary outcomes include exploring treatment effects on insomnia symptoms (Insomnia Severity Index), sleep-wake metrics from daily sleep diaries, sleep quality, fatigue, mood (depression and anxiety symptoms), and overall acceptability of the intervention.

Participants in the SleepFix intervention group will be invited to take part in a brief post-study interview exploring their experiences and acceptability with the SleepFix app and e-psychologist support.

The study will be conducted entirely online and coordinated from the Woolcock Institute of Medical Research, Sydney, Australia.

ELIGIBILITY:
Inclusion Criteria:

* 16 -24 years old
* Able to give informed online consent and if younger <18years old guardian/parental consent
* Insomnia Severity Index ≥ 10
* English fluency
* Access to a smartphone and willingness to use a mobile app for healthcare

Exclusion Criteria:

* Shift-workers with regular shifts between the hours of 8pm and 8am.
* Recent travel to a destination with >2 hours time difference (within last 7-days and with subjective reports that they are not experiencing jet lag).
* Serious medical and/or psychiatric illnesses/disorders (e.g., Epilepsy or other seizure disorders, heart failure, bipolar disorder, schizophrenia, Major Depressive disorder)
* Self-reported/diagnosed sleep disorders other than insomnia (e.g. - Obstructive Sleep Apnoea, REM/NREM sleep disorders, Restless Leg Syndrome, Narcolepsy, free running cycle & Circadian rhythm disorder)
* Currently receiving or previously received (within the last 12 months) psychotherapy for insomnia including Cognitive Behavioural Therapy (CBT).
* Pregnant
* Professional driver or operate heavy machinery

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
1. Feasibility measure: Trial efficiency data | Baseline (Week 0)
  To evaluate feasibility based on trial efficiency. Data will be assessed by:
  1. the proportion of participants who are issued an online pre-screening number and then meet criteria for telephone screening;
  2. the proportion of participants who are issued a telephone screening number indicating eligibility and then provide consent;
  3. the proportion of participants who provide consent and then are randomised into the trial.
2. Feasibility measure: Intervention uptake | 6 weeks
  To evaluate feasibility based on Intervention uptake. Data will be assessed by:
  a. the proportion of participants randomised to SleepFix intervention group who download the SleepFix app and then enter personalised data to obtain a prescribed sleep restriction window.
Feasibility measure: Data Completion of Insomnia Severity Index | Week 6 and Week 14
  The Insomnia Severity Index (ISI) is a 7-item questionnaire used to examine overall insomnia severity. It consists of a five-point Likert type scale for each item (ranging from "no problem" = 0 to "severe problem" = 4) regarding symptoms over the past 2 weeks. All items are summed with total scores ranging from 0-28. Higher scores indicate more severe insomnia.
  The investigators will count the proportion of participants randomised that successfully complete the ISI at Week 6 and Week 14 (this is two outcomes).

SECONDARY OUTCOMES:
Effects of the SleepFix intervention on ISI scores | Week 6 and Week 14
  The Insomnia Severity Index (ISI) is a 7-item questionnaire used to examine overall insomnia severity. It consists of a five-point Likert type scale for each item (ranging from "no problem" = 0 to "severe problem" = 4) regarding symptoms over the past 2 weeks. All items are summed with total scores ranging from 0-28. Higher scores indicate more severe insomnia.
  The investigators will compare the ISI in points between the SleepFix intervention group and the Sleep health control group at 6 and 14 Weeks. The investigators will also use baseline value of ISI scores in the model. Both 6 and 14 week comparisons will use a critical P-value of 0.05.
Assessing data completeness: 7-day sleep diaries | Week 6 and week 14
  To assess data completeness we will calculate the
  a. Percentage of participants that were randomised and completed their 7-day sleep diary at week 6 and week 14
  Completeness of the 7-day sleep diary will be determined by the principal investigator who will individually look at each participant's 7- day sleep diary and make a clinical judgement call whether there is enough data to assess SOL, SE, TST and WASO to be determined complete.
Assessing data completeness: Brief Pittsburgh Sleep Quality Index (B-PSQI) | Week 6 and Week 14
  Description: To assess data completeness by reporting the percentage of completed questionnaires at week 6 and week 14. Specifically, the investigators will evaluate the percentage of participants who were randomised and completed the B-PSQI questionnaire at week 6 and week 14.
Assessing data completeness: The Flinders Fatigue Scale (FFS) | Week 6 and Week 14
  Description: To assess data completeness by reporting the percentage of completed questionnaires at week 6 and week 14. Specifically, the investigators will evaluate the percentage of participants who were randomised and completed the FSS questionnaire at week 6 and week 14.
Assessing data completeness: Patient Health Questionnaire-2 (PHQ-2) | Week 6 and Week 14
  Description: To assess data completeness by reporting the percentage of completed questionnaires at week 6 and week 14. Specifically, the investigators will evaluate the percentage of participants who were randomised and completed the PHQ-2 questionnaire at week 6 and week 14.
Assessing data completeness: Generalised Anxiety Disorder Scale-2 (GAD-2) | Week 6 and Week 14
  Description: To assess data completeness by reporting the percentage of completed questionnaires at week 6 and week 14. Specifically, the investigators will evaluate the percentage of participants who were randomised and completed the GAD-2 questionnaire at week 6 and week 14.
Sleep Onset Latency (SOL) | baseline, week 6 and week 14
  Definition: The amount of time (in minutes) it takes a participant to fall asleep after attempting to sleep, as recorded in the online 7-day sleep diary.
  Reporting: We will report the mean and 95% CI (if appropriate) from both the SleepFix intervention group and Sleep health education control group.
  We will not formally statistically test treatment differences for this variable or report P-values.
Wake After Sleep Onset (WASO) | Baseline, week 6, and week 14
  Definition: The total amount of time (in minutes) a participant spends awake after initially falling asleep and before final morning awakening, as recorded in the online 7-day sleep diary.
  Reporting: We will report the mean and 95% CI (if appropriate) from both the SleepFix intervention group and Sleep health education control group.
  We will not formally statistically test treatment differences for this variable or report P-values.
Total Sleep Time (TST) | Baseline, Week 6 and Week 14
  Definition: The total amount of time (in minutes) a participant spends asleep during the night, excluding periods of wakefulness, as recorded in the online 7-day sleep diary.
  Reporting: We will report the mean and 95% CI (if appropriate) from both the SleepFix intervention group and the Sleep health education control group.
  We will not formally statistically test treatment differences for this variable or report P-values.
Sleep Efficiency (SE) | Baseline, Week 6 and Week 14
  Definition: The percentage of time spent asleep relative to total time spent in bed, calculated as (Total Sleep Time ÷ Time in Bed) × 100, as recorded in the online 7-day sleep diary.
  Reporting: We will report the mean and 95% CI (if appropriate) from both the SleepFix intervention group and the Sleep health education control group.
  We will not formally statistically test treatment differences for this variable or report P-values.
Brief Pittsburgh Sleep Quality Index (B-PSQI) | Baseline, Week 6 and Week 14
  Definition: The Brief Pittsburgh Sleep Quality Index (B-PSQI) is a 6-item self-reported questionnaire which assesses sleep quality and disturbances during the past month. The B-PSQI is derived from the original 19-item PSQI and includes items that capture key dimensions of sleep such as sleep duration, sleep latency, and sleep disturbances. Each item is scored on a 4-point Likert-type scale ranging from 0 (no difficulty) to 3 (severe difficulty), with total scores ranging from 0 to 18. Higher scores reflect poorer sleep quality.
  Reporting: The investigators will report the mean and 95% CI (if appropriate) from both the SleepFix intervention group and the Sleep Health education control group.
  The investigators will not formally statistically test treatment differences for this variable or report P-values.
The Flinders Fatigue Scale (FFS) | Baseline, Week 6 and Week 14
  Definition: The Flinders Fatigue Scale (FFS) is a 7-item self-reported instrument designed to measure the level of subjective daytime fatigue experienced over the previous two weeks. Six items consist of a 5-point Likert type scale ranging from "not at all" = 0 to "extremely" = 4. Item 5 uses a multiple-item checklist and is scored as a sum. All items are summed with total scores ranging from 0-31 with higher scores reflecting greater fatigue.
  Reporting: The investigators will report the mean and 95% CI (if appropriate) from both the SleepFix intervention group and the Sleep health education control group.
  The investigators will not formally statistically test treatment differences for this variable or report P-values.
Patient Health Questionnaire-2 (PHQ-2) | Baseline, Week 6 and Week 14
  Definition: The Patient Health Questionnaire-2 (PHQ-2) is a 2-item self-reported measure of depressive symptoms over the past 2 weeks. Participants are asked to answer questions about the severity of depressive symptoms. Scores for each question (Likert type scale "not at all" = 0 to "nearly every day" = 3) sum to a total score of 0 to 6, with higher scores indicating more severe symptoms of depression.
  Reporting: The investigators will report the median and interquartile range (IQR) from both the SleepFix intervention group and the Sleep health education control group.
  The investigators will not formally statistically test treatment differences for this variable or report P-values.
Generalised Anxiety Disorder Scale-2 (GAD-2) | Baseline, Week 6 and Week 14
  Definition: The GAD-2 is a 2-item self-reported measure of anxiety symptoms and asks how often participants have experienced anxiety symptoms in the previous two weeks. GAD-2 consists of a three-point Likert type scale for each item (ranging from "not at all" = 0 to "nearly every day" = 3). Scores for each question (Likert type scale "not at all" = 0 to "nearly every day" = 3) sum to a total score of 0 to 6. Higher scores indicate greater severity of anxiety symptoms.
  Reporting: The investigators will report the median and interquartile range (IQR) from both the SleepFix intervention group and the Sleep Health education control group.
  The investigators will not formally statistically test treatment differences for this variable or report P-values.
Acceptability of SleepFix app and e-psychologist support | Week 14
  Acceptability will be assessed through a 20-minute post-study semi-structured telephone interview (Intervention group only). Participants will be interviewed individually over the phone with the purpose of exploring their user experiences, acceptability of the sleep program and to probe their attitudes towards SleepFix integrated with e-psychologist support.
  Qualitative semi-structured interview data on user experience and acceptability of the SleepFix intervention will be analysed using thematic analysis within a framework approach. Transcripts from recordings will be read in full, coded inductively and deductively, and organised into themes that capture patterns of meaning across participants. Analysis will follow Braun and Clarke's (2006) six phases of thematic analysis including familiarisation, coding, generating themes, reviewing themes, defining/naming themes, and reporting. Representative participant quotes will be used to illustrate themes were relevant.

OTHER OUTCOMES:
Number e-psychologist support calls accessed | Week 6
  Participants in the SleepFix treatment group can access an e-psychologist support call each week during the 6 week intervention period. A minimum of 0 and a maximum of 6 e-psychologist support calls can be accessed during the intervention. The investigators will report the number of e-psychologist support calls completed from participants in the SleepFix intervention group. Reporting: this will be reported as a median and IQR.

CONTACTS AND LOCATIONS:
Overall Officials: Professor Delwyn Bartlett, Principal Investigator — Woolcock Institute of Medical Research

IPD SHARING:
Plan to Share IPD: No
The trial investigators will be given access to the cleaned data set. The project data set will be housed online in the study web portal created for the study, and all data will be password protected. To ensure confidentiality, data dispersed to project team members will be blinded of any identifying participant information.
  Data will not be shared without permission of Principal Investigators. All data available for sharing will be stored on a web-based database located in Australia. After the study, a non-identified dataset may be made available online in a data repository.

REFERENCES:
- [Background] Aji M, Glozier N, Bartlett DJ, Grunstein RR, Calvo RA, Marshall NS, White DP, Gordon C. The Effectiveness of Digital Insomnia Treatment with Adjunctive Wearable Technology: A Pilot Randomized Controlled Trial. Behav Sleep Med. 2022 Sep-Oct;20(5):570-583. doi: 10.1080/15402002.2021.1967157. Epub 2021 Aug 20. PMID 34415819
- [Background] Gordon CJ, Cheung JMY, Schrire ZM, Rahimi M, Aji M, Salomon H, Doggett I, Glozier N, Wong KKH, Marshall NS, Bartlett DJ, Grunstein RR. Integrating digital behavioural therapy for insomnia into primary care: A feasibility mixed-methods study. J Sleep Res. 2025 Jun;34(3):e14401. doi: 10.1111/jsr.14401. Epub 2024 Nov 12. PMID 39533507
- [Background] Morin CM, Belleville G, Belanger L, Ivers H. The Insomnia Severity Index: psychometric indicators to detect insomnia cases and evaluate treatment response. Sleep. 2011 May 1;34(5):601-8. doi: 10.1093/sleep/34.5.601. PMID 21532953
- [Background] Gradisar M, Lack L, Richards H, Harris J, Gallasch J, Boundy M, Johnston A. The Flinders Fatigue Scale: preliminary psychometric properties and clinical sensitivity of a new scale for measuring daytime fatigue associated with insomnia. J Clin Sleep Med. 2007 Dec 15;3(7):722-8. PMID 18198807
- [Background] Lowe B, Kroenke K, Grafe K. Detecting and monitoring depression with a two-item questionnaire (PHQ-2). J Psychosom Res. 2005 Feb;58(2):163-71. doi: 10.1016/j.jpsychores.2004.09.006. PMID 15820844
- [Background] Kroenke K, Spitzer RL, Williams JB, Monahan PO, Lowe B. Anxiety disorders in primary care: prevalence, impairment, comorbidity, and detection. Ann Intern Med. 2007 Mar 6;146(5):317-25. doi: 10.7326/0003-4819-146-5-200703060-00004. PMID 17339617
- [Background] Sancho-Domingo C, Carballo JL, Coloma-Carmona A, Buysse DJ. Brief version of the Pittsburgh Sleep Quality Index (B-PSQI) and measurement invariance across gender and age in a population-based sample. Psychol Assess. 2021 Feb;33(2):111-121. doi: 10.1037/pas0000959. Epub 2020 Oct 29. PMID 33119375
- [Background] Galgut Y, Hoyos C, Kempler L, Aji M, Grunstein RR, Gordon CJ, Bartlett DJ. Cognitive and behavioural therapy for insomnia in the treatment of adolescent insomnia: A systematic review and meta-analysis of randomised controlled trials. J Sleep Res. 2025 Aug;34(4):e14442. doi: 10.1111/jsr.14442. Epub 2024 Dec 16. PMID 39680961